CLINICAL TRIAL: NCT03671902
Title: Noninvasive Monitoring in Lower Body Negative and Positive Pressure Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James C. Leiter, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00030287 DF18055
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhage
Keywords: Phonocardiogram
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lower Body Negative/Positive Pressure (Other)
  Interventions: Device: Fluid shift

INTERVENTIONS:
Device: Fluid shift — We are using lower body negative and positive pressure to create a fluid shift in the body. This study is investigating if there are changes in phonocardiographic parameters related to changes in blood volume caused by this fluid shift

SUMMARY:
The goal of these studies is to assess the use of phonocardiograhy to monitor blood volume. We will evaluate phonocardiographic parameters in normal subjects in increasing levels of lower body negative pressure (LBNP) and lower body positive pressure (LBPP).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Good health
* Free of systemic diseases
* No contraindications to LBNP/LBPP exposure
* Normal resting systolic blood pressure (SBP, 100-140 mm Hg) and diastolic blood pressure (DBP, 60-90 mm Hg)

Exclusion Criteria:

* Pregnancy
* Prior history of cardiovascular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in the phonocardiographic systolic index (PSI) | Baseline, and at each incremental change of 5-10 mmHg up to 40 mm Hg. Total duration per arm is up to 45 min
  Measuring changes in phonocardiographic parameters related to changes in blood volume

CONTACTS AND LOCATIONS:
Overall Officials: Jay C. Buckey, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No